CLINICAL TRIAL: NCT05795062
Title: Post-Discharge Treatment Patterns and Outcomes in Patients With Venous Thromboembolism
Brief Title: Treatment Patterns Among Patients With Venous Thromboembolism in the United States
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: B0661190
Record Dates: First submitted 2023-03-06; First posted 2023-04-03 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-09

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — apixaban; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- apixaban: Patients treated with apixaban
  Interventions: Drug: apixaban
- warfarin: patients treated with warfarin
  Interventions: Drug: warfarin

INTERVENTIONS:
Drug: apixaban — patients treated with apixaban
  Groups: apixaban
Drug: warfarin — patients treated with warfarin
  Groups: warfarin

SUMMARY:
The purpose of this study is to assess outpatient treatment patterns following hospitalization for venous thromboembolism (VTE). VTE is a condition that occurs when blood clot forms in the vein.

This is a retrospective study (assessments on events that have already occurred) of healthcare claims from databases. The study sponsors will assess healthcare claim records of patients treated with either apixaban or warfarin. Assessment includes treatment persistence, switch, and stopping therapy, along with recurrent VTE and bleeding.

ELIGIBILITY:
Inclusion Criteria:

* inpatient hospitalization with primary discharge diagnosis of venous thromboembolism (VTE) (this is the index hospitalization)
* treatment with apixaban or warfarin during the hospitalization
* at least 18 years of age

Exclusion Criteria:

* Hospitalization for VTE within 6 months prior to the index hospitalization
* Diagnosis of atrial fibrillation/flutter or procedure for mechanical heart valve in the 6 months prior to the index hospitalization
* Procedure for inferior vena cava filter or diagnosis of pregnancy during the study period
* Prior use of oral anticoagulants or parenteral anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are hospitalized for venous thromboembolism (VTE) and treated with apixaban or warfarin during the hospitalization. Patients will be identified through linkage of IQVIA's hospital charge data master database (CDM) with outpatient professional fee medical claims (Dx) and longitudinal prescription claims (LRx) databases during the period of July 2018 and August 2022.
Sampling Method: Non-Probability Sample
Enrollment: 13945 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B0661190

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of eligible participants, who had hospitalization for primary diagnosis of venous thromboembolism (VTE) and received apixaban or warfarin, was extracted from databases and health claim records from 01 July 2017 to 31 December 2022 (study data identification duration of 5.5 years).
Pre-assignment Details: It is a retrospective population-based register study. Available data from eligible participants was evaluated in approximately 7 months of this retrospective, observational study per its objectives.
Groups:
- Apixaban: Participants who received apixaban (per clinical practice) during the hospitalization for primary diagnosis of VTE were included. Available data was evaluated in approximately 7 months of this retrospective, observational study.
- Warfarin: Participants who received warfarin (per clinical practice) during the hospitalization for primary diagnosis of VTE were included. Available data was evaluated in approximately 7 months of this retrospective, observational study.
Period: Overall Study
Arm/Group | Apixaban | Warfarin
Started | 11966 | 1979
Completed | 11966 | 1979
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible participants whose data was extracted and evaluated in this study and was evaluable for analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Apixaban | Warfarin | Total
Number analyzed (Participants) | 11966 | 1979 | 13945
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4737 | 878 | 5615
  >=65 years | 7229 | 1101 | 8330
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6714 | 1130 | 7844
  Male | 5252 | 849 | 6101
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Continued Treatment With Apixaban or Warfarin Following Discharge From the Hospital
Description: Following discharge from inpatient hospitalization, participants who continued apixaban or warfarin, respectively, in the outpatient setting (with outpatient treatment claim occurring on or within 30-days following the hospital discharge date) were identified.
Time Frame: From hospital discharge date through 30 days following discharge date (from the data retrieved for 5.5 years and retrospective data evaluated in approximately 7 months of this study)
Population: Eligible participants whose data was extracted and evaluated in this study and was evaluable for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 11966 | 1979
Participants | 11966 | 1979

2. Primary Outcome: Mean Number of Persistent Days
Description: Persistent days was defined as the number of days from the index date until the first of the following: treatment discontinuation, treatment switch, or the end of follow-up. Treatment index date: date of first outpatient apixaban or warfarin claim.
Time Frame: From the index date until the first of treatment discontinuation, treatment switch, or the end of follow-up, whichever occurred first (data retrieved for 5.5 years and retrospective data evaluated in approximately 7 months of this study)
Population: Eligible participants whose data was extracted and evaluated in this study and was evaluable for analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 11966 | 1979
Days | 233.5 (302.9) | 242.6 (304.4)

3. Primary Outcome: Percentage of Participants Who Discontinued Index Treatment at 6 Months Post-Discharge Index Date
Description: Discontinuation was defined as greater than or equal to (>=) 30-day gap from the run-out of days supply of the treatment (post-discharge) index prescription (that is, apixaban or warfarin) to date of next claim for the respective therapy or with no other claims for the respective therapy. The date of discontinuation was last day of day's supply of the last filled prescription. Treatment index date: date of first outpatient apixaban or warfarin claim.
Time Frame: At 6 Months post-discharge index date (data retrieved for 5.5 years and retrospective data evaluated in approximately 7 months of this study)
Population: Eligible participants whose data was extracted and evaluated in this study and was evaluable for analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 11966 | 1979
Percentage of Participants | 50.5 | 52.2

4. Primary Outcome: Percentage of Participants Who Discontinued Index Treatment at 12 Months Post-Discharge Index Date
Description: Discontinuation was defined as >= 30-day gap from the run-out of days supply of the treatment (post-discharge) index prescription (that is, apixaban or warfarin) to date of next claim for the respective therapy or with no other claims for the respective therapy. The date of discontinuation was last day of day's supply of the last filled prescription. Treatment index date: date of first outpatient apixaban or warfarin claim.
Time Frame: At 12 Months post-discharge index date (data retrieved for 5.5 years and retrospective data evaluated in approximately 7 months of this study)
Population: Eligible participants whose data was extracted and evaluated in this study and was evaluable for analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 11966 | 1979
Percentage of Participants | 72.9 | 75.2

5. Primary Outcome: Percentage of Participants Who Switched From Index Treatment at 6 Months Post-Discharge Index Date
Description: Participants were considered to have switched if they filled a prescription for oral anticoagulant (OAC) other than apixaban or warfarin, respectively (identified through national drug codes [NDC] codes in longitudinal prescription claims [LRx]) or for parenteral anticoagulant (PAC) within 30 days before or after the run-out date of index treatment. The date of the switch was defined as date of the prescription of such a therapy (OAC or PAC). Treatment index date: date of first outpatient apixaban or warfarin claim.
Time Frame: as for outcome 3
Population: Eligible participants whose data was extracted and evaluated in this study and was evaluable for analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 11966 | 1979
Percentage of Participants | 6.0 | 20.9

6. Primary Outcome: Percentage of Participants Who Switched From Index Treatment at Month 12 Post-Discharge Index Date
Description: Participants were considered to have switched if they filled a prescription for OAC other than apixaban or warfarin, respectively (identified through NDC codes in LRx) or for PAC within 30 days before or after the run-out date of index treatment. The date of the switch was defined as date of the prescription of such a therapy (OAC or PAC). Treatment index date: date of first outpatient apixaban or warfarin claim.
Time Frame: as for outcome 4
Population: Eligible participants whose data was extracted and evaluated in this study and was evaluable for analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 11966 | 1979
Percentage of Participants | 7.1 | 24.3

7. Primary Outcome: Median Time to Discontinuation From the Index Treatment
Description: Time from treatment index date to discontinuation date was described in this outcome measure. Discontinuation was defined as >= 30-day gap from the run-out of days supply of the treatment (post-discharge) index prescription (that is, apixaban or warfarin) to date of next claim for the respective therapy or with no other claims for the respective therapy. The date of discontinuation was last day of day's supply of the last filled prescription. Treatment index date: date of first outpatient apixaban or warfarin claim.
Time Frame: From initiation of index treatment post-discharge till its discontinuation (data retrieved for 5.5 years and retrospective data evaluated in approximately 7 months of this study)
Population: Eligible participants whose data was extracted and evaluated in this study and was evaluable for analysis.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 11966 | 1979
Months | 5.97 [5.83 to 6.07] | 5.67 [5.17 to 6.03]

8. Primary Outcome: Median Time to Switch From the Index Treatment
Description: Time from treatment index date to treatment switch date was described in this outcome measure. Participants were considered to have switched if they filled a prescription for OAC other than apixaban or warfarin, respectively (identified through NDC codes in LRx) or for PAC within 30 days before or after the run-out date of index treatment. The date of the switch was defined as date of the prescription of such a therapy (OAC or PAC). Treatment index date: date of first outpatient apixaban or warfarin claim.
Time Frame: From initiation of index treatment post-discharge till switch (data retrieved for 5.5 years and retrospective data evaluated in approximately 7 months of this study)
Population: Eligible participants whose data was extracted and evaluated in this study and was evaluable for analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 11966 | 1979
Months | NA [NA to NA] — The median time to switch from the index treatment could not be estimated and calculated because more than half the participants did not experience a switch. | NA [NA to NA] — The median time to switch from the index treatment could not be estimated because more than half the participants did not experience a switch.

9. Secondary Outcome: Incidence Rate of Recurrent VTE Events
Description: Recurrent VTE was defined as inpatient hospitalization with a primary diagnosis of VTE occurring 7 or more days after the first hospitalization discharge date. The date of the first observed event was flagged. Incidence rate was defined as the number of events (recurrent VTE) per 100 participant years. Treatment index date: date of first outpatient apixaban or warfarin claim.
Time Frame: From first hospitalization discharge date to subsequent inpatient hospitalization for VTE (data retrieved for 5.5 years and retrospective data evaluated in approximately 7 months of this study)
Population: Eligible participants whose data was extracted and evaluated in this study and was evaluable for analysis.
Measure: Number; unit: Events per 100 participant-years
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 11966 | 1979
Events per 100 participant-years | 1.2 | 2.5

10. Secondary Outcome: Median Time to Recurrent VTE
Description: Recurrent VTE was defined as inpatient hospitalization with a primary diagnosis of VTE occurring 7 or more days after the first hospitalization discharge date. The date of the first observed event was flagged. Treatment index date: date of first outpatient apixaban or warfarin claim.
Time Frame: as for outcome 9
Population: Eligible participants whose data was extracted and evaluated in this study and was evaluable for analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 11966 | 1979
Months | NA [NA to NA] — The median time to event could not be estimated and calculated because more than half the participants did not experience recurrent VTE. | NA [NA to NA] — The median time to event could not be estimated and calculated because more than half the participants did not experience recurrent VTE.

11. Secondary Outcome: Incidence Rate of Major Bleeding Events
Description: Major bleeding was defined as inpatient hospitalization with primary diagnosis of gastro-intestinal bleeding, intracranial hemorrhage (ICH) or other major bleeding. Incidence rate was defined as the number of events (major bleeding) per 100 participant years. Treatment index date: date of first outpatient apixaban or warfarin claim.
Time Frame: From first hospitalization discharge through first major bleeding event (data retrieved for 5.5 years and retrospective data evaluated in approximately 7 months of this study)
Population: Eligible participants whose data was extracted and evaluated in this study and was evaluable for analysis.
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 11966 | 1979
Events per 100 participant-years | 1.5 [1.2 to 1.8] | 2.0 [1.3 to 2.9]

12. Secondary Outcome: Incidence Rate of Clinically Relevant Non-Major (CRNM) Bleeding Events
Description: CRNM bleeding was defined as inpatient hospitalization with a secondary diagnosis code for bleeding (without a major bleeding code in the primary position) or an outpatient encounter with a diagnosis code in any position for CRNM gastrointestinal (GI) bleeding or other non-critical types of bleeding. Incidence rate was defined as the number of events (CRNM bleeding) per 100 participant years.
Time Frame: From first hospitalization discharge through first CRNM bleeding event (data retrieved for 5.5 years and retrospective data evaluated in approximately 7 months of this study)
Population: Eligible participants whose data was extracted and evaluated in this study and was evaluable for analysis.
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 11966 | 1979
Events per 100 participant-years | 17.7 [16.7 to 18.7] | 21.3 [18.8 to 24.1]

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not collected for the study
Description: Due to non-interventional nature of the study and nature of data sources, the minimum criteria for reporting an adverse event (that is, identifiable participant, identifiable reporter, a suspect product, and event) could not be met, hence adverse events were not planned to be collected and reported.
Arm/Group | Apixaban | Warfarin
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT05795062/Prot_SAP_000.pdf